CLINICAL TRIAL: NCT06547931
Title: Retrospective Analysis of a Cohort of Duffy-null Associated Neutrophil Count (DANC) Pediatric Patients
Brief Title: Duffy-null Associated Neutrphil Count (DANC) Pediatric Patients
Acronym: DANCChildren
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Alessandra Cattaneo, Biologist, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: 0017727
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Neutropenia Autoimmune
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Duffy null neutropenic subjects: Pediatric patients sent to our laboratory for anti-neutrophil antibodies evaluation in the suspicion of immune neutropenia
  Interventions: Other: Data collection and analysis

INTERVENTIONS:
Other: Data collection and analysis — Retrospective collection of clinical and laboratory data relating to the definition of the nature of neutropenia

SUMMARY:
There are currently no clinical and laboratory data that well characterize this neutropenia associated with the Duffy-null phenotype, particularly for pediatric subjects. In particular there are no data on the frequency of immune neutropenia in DANC neutropenic pediatric subjects.

The goal of this study is to :

* define the frequency of immune neutropenia within the cohort of DANC subjects under study
* evaluate the frequency of different degrees of neutropenia (mild-moderate-severe);
* evaluate the possible association between different degrees of neutropenia and the presence of infections.

ELIGIBILITY:
Inclusion Criteria:

* presence of Duffy-null phenotype

Exclusion Criteria:

* absence of Duffy-null phenotype

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients sent to our laboratory for the search for anti-neutrophil antibodies in the suspicion of immune neutropenia
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Immune neutropenia and DANC | Through study completion, an average of 1 year
  Frequency of immune neutropenia, expressed as the percentage of DANC subjects testing positive for anti-neutrophil antibodies out of the total DANC subjects included in the study.

SECONDARY OUTCOMES:
Distribution of mild, moderate and severe neutropenia in DANC children | Through study completion, an average of 1 year
  Frequencies in percentage of mild (1000-1500 neutrophils/ul), moderate (500-1000 neutrophils/ul) and severe (<500 neutrophils/ul) neutropenia within the DANC cohort under study

OTHER OUTCOMES:
Neutropenia severity and infections | Through study completion, an average of 1 year
  Correlation between the severity of neutropenia and the presence of infections.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggioe Policlinico, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: Yes
The data will be made public anonymously and presented as required in aggregate mode
Time Frame: Starting 6 months after publication

REFERENCES:
- [Background] Hsieh MM, Everhart JE, Byrd-Holt DD, Tisdale JF, Rodgers GP. Prevalence of neutropenia in the U.S. population: age, sex, smoking status, and ethnic differences. Ann Intern Med. 2007 Apr 3;146(7):486-92. doi: 10.7326/0003-4819-146-7-200704030-00004. PMID 17404350
- [Background] Ortiz MV, Meier ER, Hsieh MM. Identification and Clinical Characterization of Children With Benign Ethnic Neutropenia. J Pediatr Hematol Oncol. 2016 Apr;38(3):e140-3. doi: 10.1097/MPH.0000000000000528. PMID 26925714
- [Background] Rappoport N, Simon AJ, Amariglio N, Rechavi G. The Duffy antigen receptor for chemokines, ACKR1,- 'Jeanne DARC' of benign neutropenia. Br J Haematol. 2019 Feb;184(4):497-507. doi: 10.1111/bjh.15730. Epub 2018 Dec 27. PMID 30592023
- [Background] Merz LE, Li SH, Ney G, Michniacki TF, Hannibal MC, Walkovich KJ. Absolute neutrophil count nadir in healthy pediatric patients with the Duffy-null phenotype. Blood Adv. 2023 Aug 8;7(15):4182-4185. doi: 10.1182/bloodadvances.2023010368. No abstract available. PMID 37285802
- [Background] Bux J, Behrens G, Jaeger G, Welte K. Diagnosis and clinical course of autoimmune neutropenia in infancy: analysis of 240 cases. Blood. 1998 Jan 1;91(1):181-6. PMID 9414283